CLINICAL TRIAL: NCT01544088
Title: Group CBT for Chronic PTSD: RCT With Veterans
Brief Title: Group Treatment for PTSD: A Randomized Clinical Trial With Veterans
Acronym: GCBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-015-11F; 1I01CX000467-01A1 (NIH)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: PTSD
Keywords: randomized controlled trial; PTSD; cognitive behavioral treatment; group treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: GCBT (Experimental): Group Cognitive Behavioral treatment (GCBT)
  Interventions: Behavioral: Group Cognitive Behavioral Treatment (GCBT)
- Arm 2: Group Treatment (Active Comparator): Present Centered Group Treatment
  Interventions: Behavioral: Present Centered Group Treatment

INTERVENTIONS:
Behavioral: Group Cognitive Behavioral Treatment (GCBT) — GCBT is a 14 week intervention that includes components of exposure (imaginal and in vivo), cognitive restructuring, and relapse prevention.
  Arms: Arm 1: GCBT
Behavioral: Present Centered Group Treatment — The active comparison treatment is a 14 week treatment that focuses on here and now problems, especially problem solving skills concerning ongoing stressors.
  Arms: Arm 2: Group Treatment

SUMMARY:
The purpose of this study is to examine whether group cognitive behavioral treatment (GCBT) is efficacious in the treatment of PTSD in a sample of male Veterans. Veterans with a primary diagnosis of chronic PTSD will be randomly assigned to either GCBT or a supportive group treatment condition. Both treatments will consist of 14, weekly sessions. Assessment of PTSD and related symptoms will be conducted at pre-treatment, mid treatment, post-treatment, and 3-, 6-, - and 12-month follow-up.

DETAILED DESCRIPTION:
The mental health needs of Veterans within the VA Healthcare system are notable. With the substantial increase over the past 10 years in Veterans seeking Posttraumatic Stress Disorder (PTSD) treatment services, the VA system is straining to accommodate these needs, relying heavily on group-based treatments. The proposed research will take the next step in the literature on group psychotherapy for PTSD by examining a group cognitive behavioral treatment (GCBT) program with promising pilot data. This application supports a randomized controlled trial, which will compare GCBT with Supportive Group Psychotherapy (SGP). The trial will involve 196 male Veterans with combat-related PTSD who will be randomly assigned to GCBT (n= 98) or SGP (n =98) to determine efficacy within a naturalistic care environment. Outcome data will be collected pre-treatment, mid-treatment, post-treatment, and 3-, 6- and 12-month follow-up. Two aims are included, one focusing on outcome with respect to PTSD symptom severity, the second focusing on treatment generalization to comorbid emotional disorders (major depressive disorder, generalized anxiety disorder, and alcohol abuse), and distress and impairment. Data will be examined using latent growth curve modeling, with emphasis on determining efficacy and effectiveness. The information provided by the proposed project could assist in developing more effective care models for individuals with chronic PTSD from numerous traumatic experiences. Additionally, this project represents an effort to move the literature on group-based treatments for PTSD ahead, through inclusion of advanced methodological and analytic approaches.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of DSM-IV (American Psychiatric Association, 2000) criteria for chronic, PTSD (symptoms lasting 3 months or more)
* male, Veteran
* be free of psychosis and impaired cognitive function caused by traumatic brain injury or dementia

Exclusion Criteria:

* a current diagnosis of substance dependence or unstable bipolar disorder
* currently involved in psychosocial treatment for PTSD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Sloan, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through Freedom of Information Act.

REFERENCES:
- [Background] Sloan DM, Unger W, Lee DJ, Beck JG. A Randomized Controlled Trial of Group Cognitive Behavioral Treatment for Veterans Diagnosed With Chronic Posttraumatic Stress Disorder. J Trauma Stress. 2018 Dec;31(6):886-898. doi: 10.1002/jts.22338. Epub 2018 Nov 29. PMID 30499227
- [Background] Sloan DM, Unger W, Gayle Beck J. Cognitive-behavioral group treatment for veterans diagnosed with PTSD: Design of a hybrid efficacy-effectiveness clinical trial. Contemp Clin Trials. 2016 Mar;47:123-30. doi: 10.1016/j.cct.2015.12.016. Epub 2015 Dec 21. PMID 26718094
- [Derived] Marx BP, Lee DJ, Norman SB, Bovin MJ, Sloan DM, Weathers FW, Keane TM, Schnurr PP. Reliable and clinically significant change in the clinician-administered PTSD Scale for DSM-5 and PTSD Checklist for DSM-5 among male veterans. Psychol Assess. 2022 Feb;34(2):197-203. doi: 10.1037/pas0001098. Epub 2021 Dec 23. PMID 34941354

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
Started | 98 | 100
Completed | 61 | 79
Not Completed | 37 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment | Total
Number analyzed (Participants) | 98 | 100 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 67 | 142
  >=65 years | 23 | 33 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.40 (11.44) | 57.22 (12.51) | 55.82 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 98 | 100 | 198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 19 | 33
  White | 75 | 72 | 147
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 100 | 198
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — Total score range = 0-80; higher scores indicate greater symptom severity
  units on a scale | 39.84 (9.84) | 39.37 (9.52) | 39.60 (9.66)
Beck Depression Inventory, II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — Total score range = 0-63; higher scores indicate greater symptom severity
  units on a scale | 23.85 (11.95) | 23.94 (11.65) | 23.89 (11.77)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — Total score range = 0-63; higher scores indicate greater symptom severity
  units on a scale | 18.22 (11.31) | 20.97 (12.15) | 19.61 (11.80)
Short-Form Health Survey (SF-36) [Mean (Standard Deviation); unit: units on a scale] — Total score range = 0-200; higher scores indicate greater functioning
  units on a scale | 39.43 (26.60) | 42.88 (26.37) | 41.18 (26.47)

OUTCOME MEASURES:

1. Primary Outcome: Clinician-Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The CAPS-5 is a semi-structured interview to assess presence and severity of PTSD symptoms. The total score on the CAPS will be used as the primary outcome measure in this study. Total score range = 0-80; higher scores indicate greater symptom severity.
Time Frame: 12 months
Population: Primary treatment outcomes were examined using hierarchical linear modeling.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
Number analyzed (Participants) | 98 | 100
units on a scale | 28.76 (13.46) | 31.87 (14.70)

2. Secondary Outcome: Beck Depression Inventory, II (BDI-II)
Description: The BDI is a self-report inventory that indexes depression symptom severity. Total score range = 0-63; higher scores indicate greater symptom severity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
Number analyzed (Participants) | 98 | 100
units on a scale | 18.95 (12.67) | 22.29 (13.20)

3. Secondary Outcome: Short-Form Health Survey (SF-36)
Description: The SF-36 is a measure of functional impairment. Total score range = 0-200; higher scores indicate greater functioning.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
Number analyzed (Participants) | 98 | 100
units on a scale | 55.00 (28.71) | 59.05 (27.21)

4. Secondary Outcome: Beck Anxiety Inventory (BAI)
Description: The BAI is a self-report measure of general anxiety symptom severity. Total score range = 0-63; higher scores indicate greater symptom severity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
Number analyzed (Participants) | 98 | 100
units on a scale | 15.23 (12.34) | 18.67 (13.77)

ADVERSE EVENTS:
Time Frame: 1 year, 4 months
Description: Adverse events were collected based on participant self-report as well as documentation in the VA electronic medical record. As standard practice, all adverse reports were documented, whether or not they were probably or likely related to study participation.
Arm/Group | Group Cognitive Behavioral Treatment (GCBT) | Present Centered Group Treatment
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/100
Serious Adverse Events (participants affected / at risk) | 15/98 | 22/100
Other Adverse Events (participants affected / at risk) | 0/98 | 0/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Cognitive Behavioral Treatment (GCBT) (N=98) | Present Centered Group Treatment (N=100)
hospitalization due to medical illness (Surgical and medical procedures) | 2 (2) | 4 (4) — Medical hospitalization due to medical/surgical procedures
psychiatric hospitalization (Psychiatric disorders) | 4 (4) | 9 (9) — hospitalization for substance-use related disorder, a condition that predated study entry. Moreover, hospitalization occurred during the follow up assessment phase of the study.
General disorders (General disorders) | 2 (2) | 4 (4) — hospitalization for general disorders
Uninary disorder (Renal and urinary disorders) | 1 (1) | 2 (2) — hospitalization due to renal or urinary disorder
Infection disease (Infections and infestations) | 3 (3) | 2 (2) — hospitalization due to infectious disease
GI illness (Gastrointestinal disorders) | 3 (3) | 1 (1) — hospitalization due to GI disorders

LIMITATIONS AND CAVEATS:
No women veterans were included in the study, therefore findings are not generalizable to women veterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-28): https://cdn.clinicaltrials.gov/large-docs/88/NCT01544088/Prot_SAP_000.pdf